CLINICAL TRIAL: NCT06637150
Title: A Phase III Randomized Controlled Trial Comparing Dalpicilib-Enhanced Adjuvant Endocrine Therapy with Standard Adjuvant Endocrine Therapy in ER+ HER2- Lymph Node-Negative Early Breast Cancer with Risk Factors
Brief Title: Dalpicilib-Enhanced Vs. Standard Endocrine Therapy in ER+ HER2- Early Breast Cancer
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N081
Record Dates: First submitted 2024-09-28; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- standard endocrine therapy (Active Comparator): standard endocrine therapy
  Interventions: Drug: endocrine therapy
- standard endocrine therapy plus dalpicilib (Experimental): standard endocrine therapy plus dalpicilib
  Interventions: Drug: Dalpicilib; Drug: endocrine therapy

INTERVENTIONS:
Drug: Dalpicilib — Dalpicilib 100 mg once daily from day 1 to day 21, every 4 weeks, for a total of 3 years, in combination with endocrine therapy for 5 years.
  Arms: standard endocrine therapy plus dalpicilib
Drug: endocrine therapy — standard endocrine therapy

SUMMARY:
This study aims to conduct a randomized controlled clinical trial to compare the efficacy and safety of dalpicilib combined with endocrine therapy versus standard endocrine therapy in ER-positive, HER2-negative, lymph node-negative patients with risk factors, in order to further optimize the regimen for adjuvant endocrine therapy in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18-70 years
2. ECOG score of 0-1
3. Histologically confirmed unilateral invasive cancer (regardless of pathology type)
4. No macroscopic or microscopic tumor residue after surgical resection
5. Early-stage breast cancer, pathologically confirmed as ER-positive and HER2-negative (ER-positive defined as immunohistochemical detection of ER >10% of tumor cells positive; HER2 0-1+ or HER2 2+ but FISH negative, with no amplification, defined as HER2-negative)
6. Postoperative pathological staging of pT1c or above, N0M0, and meeting one of the following criteria: (1) G3; (2) G2 and meeting one of the following: i. Ki-67 ≥20%; ii. 21-gene recurrence score ≥26 or high genomic risk profile; iii. Age ≤40 years and vascular invasion positive
7. No prior neoadjuvant treatment
8. Time from surgery or completion of chemotherapy or radiotherapy (whichever occurs later) to randomization does not exceed 8 weeks
9. Good postoperative recovery, at least 1 week after surgery
10. Normal function of major organs, meeting the following criteria: (1) Hematological criteria: HB ≥90 g/L (no blood transfusion in the last 14 days); ANC ≥1.5 × 10^9 /L; PLT ≥100 × 10^9 /L; (2) Biochemical criteria: TBIL ≤1.5 × ULN (upper limit of normal); ALT and AST ≤3 × ULN; serum Cr ≤1.5 × ULN
11. Women of childbearing age must use contraception during treatment
12. Subjects voluntarily join this study, sign informed consent, demonstrate good compliance, and cooperate with follow-up

Exclusion Criteria:

1. Bilateral breast cancer or ductal/lobular carcinoma in situ (DCIS/LCIS)
2. Received treatment for advanced disease
3. Metastasis at any site
4. Any tumor > T4a (with skin involvement, fixation, inflammatory breast cancer)
5. Clinically or radiologically suspected malignancy in the contralateral breast not confirmed and requiring biopsy
6. Received neoadjuvant therapy, including chemotherapy, radiotherapy, and endocrine therapy
7. History of malignant tumors within the past 5 years (excluding basal cell carcinoma of the skin and cervical carcinoma in situ), including contralateral breast cancer
8. Patient has been enrolled in other clinical trials
9. Patient has severe systemic diseases and/or uncontrolled infections that prevent participation in the study
10. Severe cardiovascular or cerebrovascular diseases within 6 months prior to randomization (e.g., unstable angina, chronic heart failure, uncontrolled hypertension >150/90 mmHg, myocardial infarction, or stroke)
11. Known allergy to relevant medications
12. Women of childbearing age who refuse contraception during treatment and for 8 weeks after treatment completion
13. Pregnant or breastfeeding women
14. Positive pregnancy test before drug administration after joining the trial
15. Individuals with mental illness or cognitive impairment who cannot understand the trial protocol and its side effects, unable to comply with the protocol and follow-up (systematic assessment required prior to enrollment)
16. Individuals without personal freedom and independent civil capacity

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 1388 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2030-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
Invasive Disease Free Survival | From enrollment to 3 years post-treatment
  Invasive Disease Free Survival

SECONDARY OUTCOMES:
3-Year Disease-Free Survival | From enrollment to 3 years post-treatment
Overall Survival | From enrollment to 3 years post-treatment
  Overall Survival
safety | From enrollment to 3 years post-treatment
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Patient reported outcomes | From enrollment to 3 years post-treatment
  Patient-Reported Outcomes (PROs) Assessed by the EORTC QLQ-C30 Questionnaire. Provide a brief description of what aspects of the patient's health or experience the tool will measure (e.g., quality of life, symptom burden, treatment side effects).

CONTACTS AND LOCATIONS:
Locations (1):
- breast cancer institute of Fudan University Cancer Hospital, shanghai, shanghai, Shanghai, China

IPD SHARING:
Plan to Share IPD: No